CLINICAL TRIAL: NCT05108389
Title: Sonoclot to Evaluate Thrombotic Risk in Proteinuric Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 19OB011
Record Dates: First submitted 2021-10-05; First posted 2021-11-04 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Pregnancy Complications; Proteinuria in Pregnancy; Chronic Kidney Diseases; Venous Thromboembolism
Keywords: Pregnancy Proteinuria Thrombosis
MeSH Terms: conditions — Pregnancy Complications; Renal Insufficiency, Chronic; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Pregnant women with kidney disease: Pregnant women with kidney disease. No intervention.
  Interventions: Diagnostic Test: Viscoelastic haemostasis monitor output

INTERVENTIONS:
Diagnostic Test: Viscoelastic haemostasis monitor output — Observational

SUMMARY:
There is a lack of consensus on whether women with proteinuric kidney disease benefit from prophylactic anticoagulation during pregnancy to reduce the risk of venous thromboembolism.

This pilot study will investigate the feasibility of obtaining thrombosis profile data using a viscoelastic haemostasis monitor - Sonoclot - from pregnant women with kidney disease, and exploratory analyses to elucidate correlations between output values and clinical parameters

DETAILED DESCRIPTION:
Pregnancy is a risk factor for women developing blood clots in veins (VTE). The risk is highest towards the end of pregnancy and in the few weeks following delivery. VTE can cause swollen painful legs due to clots in the deep veins (DVT) and/or blood clots in the lung vessels leading to chest pain, breathlessness and loss of blood pressure. VTE is the leading direct cause of death in pregnant women in the UK (affecting 1.4 per 100,000 pregnancies). Additional risk factors for VTE (including obesity, family history, previous history of blood clots and Caesarean section) are routinely valuated through standard care and treatment to thin blood with low molecular weight heparin (LWMH) injections is offered to those at highest risk. Women with kidney disease comprise a very small proportion of all pregnancies and are hence under-represented in large-scale studies to evaluate VTE risk.

Outside of pregnancy, patients with kidney conditions associated with heavy leakage of protein into urine through damaged microscopic filters (glomeruli) plus low blood protein plus swelling (the "nephrotic syndrome") have an increased risk of VTE. VTE risk is increased as a result of (a) concentration of blood within blood vessels due to fluid leak into tissues, (b) decreased flow of blood through veins due to circulating volume and decreased mobility and (c) an imbalanced loss of proteins in urine that favour or inhibit blood clotting. There is evidence to support blood thinning treatment to reduce the risk of VTE in patients with one cause of nephrotic syndrome - membranous nephropathy - and many clinicians choose to offer blood thinning treatment to patients with other causes of nephrotic syndrome if they believe the patient is at increased risk of clots.

There are no clinical data to confirm a benefit of blood thinning treatments to prevent VTE in pregnant women with nephrotic syndrome, but, faced with the lack of published studies, consensus guidelines published in 2018 recommend that women with nephrotic syndrome should be treated during pregnancy and for 6 weeks after birth.

There is a lack of consensus on whether women with less severe protein leak during pregnancy should be offered blood thinning injections. An international survey of clinicians caring for women with these conditions reports a wide range in practice from some offering treatment to all with a protein leak (urine protein:creatinine ratio) >100mg/mmol, to others only considering treatment if leak was >300mg/mmol AND evidence of low blood protein AND swelling.

VTE prophylaxis with LMWH is standard of care for medical in-patients and for out-patient treatment in pregnant women identified to be at increased VTE risk. Although LMWH treatment is not associated with any adverse pregnancy outcomes, it is uncomfortable, inconvenient and can interfere with delivery plans if spinal or epidural anesthetic is required.

There are, therefore, women receiving LMWH prophylaxis because of increased urine protein leak despite inadequate evidence to prove the benefit of this strategy and insufficient clinical tools to triage risk profiles for these patients.

There are no routine laboratory tests that offer a direct measurement of thrombotic risk. Sonoclot is established technology that has been utilised to quantify bleeding risk after cardiac surgery and disseminated clotting abnormalities, and adequacy of anticoagulation in haemodialysis patients and during treatment with direct acting oral anticoagulants. In addition to predicting bleeding risk, results also identify clotting risk. This has previously been studied in women taking oral contraception and in normal pregnancy with both identifying patterns consistent with increased thrombotic risk during pregnancy or with combined oral contraceptive use.

This study aims to assess the feasibility of conducting a clinical trial using Sonoclot results to identify which pregnant women with kidney disease are at increased risk of VTE and which are not, to define treatment protocols with LMWH prophlyaxis. This pilot study will assess the correlations between Sonoclot results, urine protein leak, gestational age, routine laboratory test results and routine VTE risk assessment tools.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed pregnancy by ultrasound scanning or urine or serum beta-HCG
* Chronic kidney disease stage 1 to 5, defined as abnormalities of serum creatinine, urine constituents or renal tract anatomy for more than 3 months, or genetic traits associated with renal disease

Exclusion Criteria:

* Known primary thrombophilia (including factor V Leiden, prothrombin mutations, protein C deficiency, protein S deficiency)
* Treatment with low molecular weight heparin in 24 hours prior to consent
* Suspected or confirmed active pre-eclampsia or superimposed pre-eclampsia

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women attending the combined renal-obstetric outpatient service at Nottingham University Hospitals NHS Trust, UK
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Proteinuria (log) to clot time correlation | Through study completion, an average of 9 months
  Univariate linear regression analysis of clot time vs log[urine protein:creatinine ratio]

SECONDARY OUTCOMES:
Proteinuria to clot time correlation | Through study completion, an average of 9 months
  Univariate linear regression analysis of clot time vs urine protein:creatinine ratio
Proteinuria (<>100mg/mmol) to clot time correlation | Through study completion, an average of 9 months
  Comparison of mean clot time vs urine protein:creatinine rate < or ≥ 100 mg/mmol
Proteinuria (<>300mg/mmol) to clot time correlation | Through study completion, an average of 9 months
  Comparison of mean clot time vs urine protein:creatinine rate < or ≥ 300 mg/mmol

OTHER OUTCOMES:
Exploratory | Through study completion, an average of 9 months
  Correlation of Sonoclot data with treatment options as per routine clinical care (aspirin, LMWH).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hall, MB MD FRCP, Principal Investigator — Nottingham University Hospitals
Locations (1):
- Nottingham University Hospitals, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised and aggregated data available to share with collaborators